CLINICAL TRIAL: NCT01154101
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase IIa Study of the Clinical Activity, Safety, and Tolerability of SRT2104 in Subjects With Moderate to Severe Plaque-Type Psoriasis
Brief Title: Study of the Clinical Activity, Safety, and Tolerability of SRT2104 in Subjects With Moderate to Severe Plaque-Type Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sirtris, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114296
Record Dates: First submitted 2010-04-22; First posted 2010-06-30 (Estimated); Results first posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-09

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — SRT2104

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 2 - 500mg SRT2104/placebo dose group (Active Comparator): 10 subjects will be randomized 4:1 (SRT2104: placebo) in each of 3 treatment arms (250mg, 500mg, or 1000mg).
  Cohort 2 will commence after Cohort 1 has completed 28 consecutive days of dosing, followed by the completion of a safety review by an Independent Safety Review Committee.
  Cohort 2 will be administered at approximately the same time every day, approximately 15 minutes following the consumption of food. Subjects must wait at least 1 hour after dosing before consuming additional calories. Dietary recommendations for the meal that precedes dosing will be provided to the study subjects by the clinical site staff.
  Interventions: Drug: Placebo; Drug: SRT2104
- Cohort 3 - 1000mg SRT2104/placebo dose group (Active Comparator): 10 subjects will be randomized 4:1 (SRT2104: placebo) in each of 3 treatment arms (250mg, 500mg, or 1000mg).
  Cohort 3 will commence after Cohort 2 has completed 28 consecutive days of dosing, followed by the completion of a safety review by an Independent Safety Review Committee.
  Cohort 3 will be administered four SRT2104 capsules at approximately the same time every day, approximately 15 minutes following the consumption of food. Subjects must wait at least 1 hour after dosing before consuming additional calories. Dietary recommendations for the meal that precedes dosing will be provided to the study subjects by the clinical site staff.
  Interventions: Drug: Placebo; Drug: SRT2104
- Cohort 1 - 250mg SRT2104/placebo dose group (Active Comparator): 10 subjects will be randomized 4:1 (SRT2104: placebo) in each of 3 treatment arms (250mg, 500mg, or 1000mg).
  Cohort 1 will be administered at approximately the same time every day, approximately 15 minutes following the consumption of food. Subjects must wait at least 1 hour after dosing before consuming additional calories. Dietary recommendations for the meal that precedes dosing will be provided to the study subjects by the clinical site staff.
  Dosing for Cohort 2 will not commence until Cohort 1 has completed 28 consecutive days of dosing, followed by the completion of a safety review by an Independent Safety Review Committee.
  Interventions: Drug: Placebo; Drug: SRT2104

INTERVENTIONS:
Drug: Placebo — For the placebo product, the SRT2104 drug substance will be replaced by microcrystalline cellulose (Avicel® PH 105) to match the SRT2104 investigational product.
Drug: SRT2104 — SRT2104 drug substance is a new chemical entity which is supplied as a fine, yellowish/amber powder. The SRT2104 investigational product is prepared by packing 250 mg of micronized SRT2104 powder with no additional additives into a size 00 opaque, hard gelatin capsule, packaged in dosing bottles containing a single daily dose.

SUMMARY:
This double-blind, placebo-controlled study will be conducted at 5 study centers in the United States. Approximately 30 subjects with moderate to severe plaque-type psoriasis will take part. The study will consist of a screening period of up to 21 days, a 12-week treatment period with 7 on-treatment clinic visits (approximately one every 2 weeks) and a post-dosing follow-up clinic visit approximately 30 days after the last dose of study drug is taken.

Subjects will be randomized to receive either 250mg, 500mg or 1000mg of study drug or placebo. Study drug will be taken by mouth on a full stomach, every day for 84 days.

Vital signs, clinical laboratory results (hematology, chemistry, and urinalysis), ECGs and physical examinations will be assessed at periodic intervals from Day 1 through Day 84.

A skin biopsy will be taken at the beginning and the end of the dosing period to evaluate any effects of the study drug on psoriasis. Investigators will perform other psoriasis evaluations (including the Psoriasis Area and Severity Index [PASI] and the Physician's Global Assessment [PGA] at 5 different times throughout the study to quantify the effects of SRT2104 on psoriasis activity.

Subjects will complete questionnaires throughout the study, to document their sense of well-being and mood at 4 different times during the study.

Five blood samples will be obtained at different timepoints during the study, to measure the amount of SRT2104 in the body.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent to participate in the study
* Be male or female aged 18 to 80 years (inclusive)
* Have a diagnosis of clinically confirmed, stable (without recent documented flare within 30 days prior to the Screening Visit), plaque-type psoriasis for at least 6 months involving ≥10% of body surface area
* Have a baseline PASI of ≥10
* Be a candidate for systemic psoriasis therapy, in the opinion of the investigator
* If a female subject of child-bearing potential, be willing to use reliable contraception for the duration of the study, through the 30 day safety follow up telephone call
* Be willing and able to comply with the protocol for the duration of the study

Exclusion Criteria:

* Has received systemic non-biologic psoriasis therapy or PUVA phototherapy within 4 weeks prior to the Screening Visit, or had topical psoriasis treatment or UVB phototherapy within 2 weeks prior to the Screening Visit
* Has received previous treatment with biologic agents within 5 drug half-lives (or within 3 months if half-life is unknown) prior to the first dose of SRT2104
* Has received a live vaccination within 4 weeks prior to the Screening Visit or intends to have a live vaccination during the course of the study
* Use of any other non-psoriatic prescription drug therapy, with the exception of any prescription medication administered at a stable dose for at least 6 weeks prior to the Screening Visit; however, the administration of proton pump inhibitors during the study dosing period is prohibited
* Use of any dietary or herbal supplements, with the exception of those administered at a stable dose for at least 6 weeks prior to the Screening Visit
* Has received any investigational drug or experimental procedure within 30 days prior to the first dose of SRT2104
* Has an active infection (e.g., sepsis, pneumonia, abscess, etc.) or be at high risk of developing an infection, in the opinion of the investigator, prior to the first dose of SRT2104
* Has a history of a positive tuberculosis test or a positive tuberculosis test at the Screening Visit that cannot be attributed to a prior BCG inoculation
* Has a positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of the Screening Visit
* Has a positive test for HIV antibody
* Has an abnormal chest x-ray at the Screening Visit which, in the opinion of the investigator, would preclude entry into the trial
* Has a 12-lead electrocardiogram (ECG) with changes considered to be clinically significant on medical review including prolonged QTc intervals as defined below:
* QTcB ≥450 msec (based on single or average QTc value of triplicate ECGs obtained over a brief period)
* QTcB ≥480 msec in subjects with Bundle Branch Block
* Has renal or liver impairment, defined as:
* Serum creatinine level of ≥ 1.4 mg/dL for females and ≥ 1.5 mg/dL for males
* AST and ALT ≥ 2xULN or
* Alkaline phosphatase and bilirubin > 1.5xULN (an isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%)
* Has active neoplastic disease or history of neoplastic disease within 5 years of study entry (except for basal or squamous cell carcinoma of the skin, or carcinoma in situ which have been definitively treated with standard of care approaches)
* Is pregnant or breast-feeding. Confirmation that a female subject is not pregnant must be established by negative pregnancy tests at Screening and Day 1
* Has a significant history of alcoholism or drug/chemical abuse, or consumes more than 3 standard units/day of alcohol. A standard unit of alcohol is defined as 250 mL of beer, 25 mL of spirit, or 125 mL of wine
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation
* Has an acute or chronic illness which, in the opinion of the investigator, could pose a threat or harm to the subject

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-06-07 (Actual); Primary Completion 2011-11-09 (Actual); Study Completion 2011-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (7):
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Johnston, Rhode Island
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Krueger JG, Suarez-Farinas M, Cueto I, Khacherian A, Matheson R, Parish LC, Leonardi C, Shortino D, Gupta A, Haddad J, Vlasuk GP, Jacobson EW. A Randomized, Placebo-Controlled Study of SRT2104, a SIRT1 Activator, in Patients with Moderate to Severe Psoriasis. PLoS One. 2015 Nov 10;10(11):e0142081. doi: 10.1371/journal.pone.0142081. eCollection 2015. PMID 26556603
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 114296 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114296 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114296 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114296 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114296 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114296 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 40 participants with moderate to severe plaque-type psoriasis were enrolled. This study was conducted at eight centers in the United States: New York (2); Missouri (1); Oregon (1); Pennsylvania (1); Rhode Island (1); Texas (1); Washington (1), from 07 June 2010 to 09 November 2011.
Pre-assignment Details: Participants were asked to sign the informed consent form (ICF) at the Screening Visit, which was conducted within 21 days prior to administration of the first dose of study drug on Day 1.
Groups:
- Placebo: Eligible participants received SRT2104 matching placebo capsules, orally, once daily after meal (at the same time every dosing day) for 12 weeks.
- SRT2104 0.25 g: Eligible participants received SRT2104 0.25 gram (g) capsules, orally, once daily after meal (at the same time every dosing day) for 12 weeks.
- SRT2104 0.5 g: Eligible participants received SRT2104 0.5 g capsules, orally, once daily after meal (at the same time every dosing day) for 12 weeks.
- SRT2104 1.0 g: Eligible participants received SRT2104 1.0 g capsules, orally, once daily after meal (at the same time every dosing day) for 12 weeks.
- No Treatment: Eligible participants in this arm received no treatment. No treatment arm was used when participants were randomized but discontinued prior to dosing.
Period: Overall Study
Arm/Group | Placebo | SRT2104 0.25 g | SRT2104 0.5 g | SRT2104 1.0 g | No Treatment
Started | 7 | 9 | 12 | 11 | 1
Completed | 7 | 5 | 9 | 9 | 0
Not Completed | 0 | 4 | 3 | 2 | 1
Not completed — Adverse Event | 0 | 2 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Sex and Race assessments were performed for the entire population (40 participants). However, for Age only 39 participants were available (1 participant withdrew from the study from the 'No Treatment group') and hence data was not collected for that participant.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | SRT2104 0.25 g | SRT2104 0.5 g | SRT2104 1.0 g | No Treatment | Total
Number analyzed (Participants) | 7 | 9 | 12 | 11 | 1 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: For the "no treatment" group: the single participant in this arm had withdrawn from the study, therefore the age data was not collected for this single participant in this arm.
  Years
    number analyzed (Participants) | 7 | 9 | 12 | 11 | 0 | 39
    (all) | 51.4 (14.88) | 40.6 (16.05) | 49.3 (14.41) | 44.6 (13.58) |  | 46.4 (14.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 0 | 5 | 1 | 10
  Male | 6 | 6 | 12 | 6 | 0 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 1 | 0 | 4
  White | 6 | 7 | 10 | 10 | 1 | 34
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Clinical Activity by Improvement Score (Using Krueger Criteria): Number of Participants With Good or Excellent Improvement Score Based on Histological Assessments of Skin Biopsies After 12 Weeks of Exposure
Description: According to the Krueger criteria, improvement score is classified as Good improvement defined as reduction in epidermal thickness by at least 30% normalized keratinocyte differentiation but most keratinocytes still express K16. Excellent improvement defined as reduction in epidermal thickness to normal or almost normal normalized keratinocyte differentiation and absent keratinocyte expression of K16. No improvement defined as no improvement in epidermal thickness keratinocyte differentiation or K16 expression on keratinocytes. A binomial response was defined for each participant according to whether the participant had an improvement score of "good or excellent improvement" (response=1) or not (response=0). Number of participants with good or excellent improvement score are presented.
Time Frame: 12 weeks
Population: The Efficacy Analysis Set (EAS) population comprised of all randomized participants who took at least one dose of study medication, had at least one activity measurement at Baseline, at least one post-Baseline study visit. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- SRT2104 0.25 g: Eligible participants received SRT2104 0.25 g capsules, orally, once daily after meal (at the same time every dosing day) for 12 weeks.
Arm/Group | Placebo | SRT2104 0.25 g | SRT2104 0.5 g | SRT2104 1.0 g
Number analyzed (Participants) | 7 | 6 | 9 | 11
Participants | 1 | 3 | 4 | 2

2. Primary Outcome: Number of Participants With Any Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e., lack of efficacy), abuse or misuse. SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant. The AE category in the data table includes participants who experienced serious or non-serious adverse events or both.
Time Frame: Up to Follow-up (Day 114)
Population: Safety Analysis Set (SAF) population which comprised of all participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SRT2104 0.25 g | SRT2104 0.5 g | SRT2104 1.0 g
Number analyzed (Participants) | 7 | 9 | 12 | 11
Participants
  AE | 3 | 4 | 9 | 11
  SAE | 0 | 2 | 0 | 1

3. Primary Outcome: Number of Participants With Hematology and Coagulation Abnormalities of Potential Clinical Concern
Description: Hematology parameters included hemoglobin, hematocrit, red blood cell count, red cell distribution width, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, platelets, white blood cell count and complete white blood cell count differential. Coagulation parameters included activated partial thromboplastin time and prothrombin time/international normalized ratio. The potential clinical concern range for hematology parameters were: white blood cell count (low: <0.67x10^9/Liter x lower limit of normal [LLN] and high: >1.82x10^9/L x upper limit of normal [ULN]), neutrophil count: (low: <0.83x10^9/Liter x LLN), hemoglobin (low: <0.85 gram/Liter x LLN and high: >1.03 gram/Liter x ULN for males and >1.13 gram/Liter x ULN for females), hematocrit with units ratio (high: >1.02 x ULN for males and >1.17 x ULN for females), platelet count (low: <0.67x10^9/Liter x LLN and high >1.57x10^9/Liter x ULN) and lymphocytes (low: <0.81x10^9/Liter x LLN).
Time Frame: Up to Follow-up (Day 114)
Population: SAF Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SRT2104 0.25 g | SRT2104 0.5 g | SRT2104 1.0 g
Number analyzed (Participants) | 7 | 9 | 12 | 11
Participants | 0 | 0 | 1 | 2

4. Primary Outcome: Number of Participants With Clinical Chemistry Abnormalities of Potential Clinical Importance
Description: The potential clinical concern range for clinical chemistry parameters were: Albumin:(low: <0.86 gram/Liter x LLN), Calcium:(low: <0.91 millimol/Liter [mmol/L] x LLN and high: >1.06 mmol/L x ULN), Creatinine: (high: >1.3 mmol /L x ULN), Glucose: (low: <0.71 mmol/L x LLN, high: >1.41 mmol/L x ULN), Magnesium: (low: <0.63 mmol/L x LLN, high: >1.03 mmol/L x ULN), Phosphorus: (low: <0.8 mmol/L x LLN, high: >1.14 mmol/L x ULN), Sodium: (low: <0.96 mmol/L x LLN, high: >1.03 mmol/L x ULN), Urea: (high: >1.5 mmol/L x ULN), Gamma glutamyl transferase: (high: >2 International units per L x ULN), Total bilirubin (high: 1.5 x ULN), both alanine amino transferase and aspartate amino transferase (high:≥ 2x ULN Units/L) and Bicarbonate: (low: <18 mmol/L and high: >32 mmol/L). Number of participants with clinical chemistry abnormalities of potential clinical importance are presented.
Time Frame: Up to Follow-up (Day 114)
Population: SAF Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SRT2104 0.25 g | SRT2104 0.5 g | SRT2104 1.0 g
Number analyzed (Participants) | 7 | 9 | 12 | 11
Participants | 4 | 3 | 5 | 5

5. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Values
Description: 12-lead ECG was performed in the rested state with the participant in the supine position with ECG leads on for at least 5 minutes prior to ECG recording. ECGs included PR (PQ), QRS, QT and QT corrected by Bazett's formula (QTcB), QT corrected by Fridericia's formula (QTcF) intervals. Identification of any conduction abnormalities were recorded in the eCRF. If a participant's QTc intervals were prolonged, then the ECG was done in triplicate with results reported as an average of the three ECGs. Number of participants with abnormal electrocardiogram (ECG) values are presented.
Time Frame: Up to Follow-up (Day 114)
Population: SAF Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SRT2104 0.25 g | SRT2104 0.5 g | SRT2104 1.0 g
Number analyzed (Participants) | 7 | 9 | 12 | 11
Participants | 3 | 1 | 4 | 6

6. Primary Outcome: Number of Participants With Vital Signs of Potential Clinical Importance
Description: Vital sign assessments included measurements of resting heart rate and blood pressure. Potential clinical concern range for systolic blood pressure: <85 and >160 millimeter of mercury (mmHg), for diastolic: <45 and >100 mmHg and heart rate: <40 and >110 beats per minute. Number of participants with vital signs of potential clinical importance are presented.
Time Frame: Up to Follow-up (Day 114)
Population: SAF Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SRT2104 0.25 g | SRT2104 0.5 g | SRT2104 1.0 g
Number analyzed (Participants) | 7 | 9 | 12 | 11
Participants | 0 | 0 | 0 | 2

7. Secondary Outcome: Number of Participants With Clinical Activity in Psoriasis Area and Severity Index (PASI) Score After 4, 8, and 12 Weeks of Exposure
Description: PASI score was determined by evaluation of body surface area (BSA) covered by plaque psoriasis in 4 areas (head/neck, arms, trunk and legs with area score of 0.1, 0.2, 0.3 and 0.4 respectively). This test included combination of both degree of involvement (assessed as per the % of affected body area using a 7-point scale such that 0=0% involvement, 1=1-9%, 2=10-29%, 3=30-49%, 4=50-69%, 5=70-89% and 6=90-100%) and severity (evaluated individually using a 5-point scale that ranged as 0=No evidence of sign, 1=slight evidence, 2=moderate evidence, 3=marked evidence and 4=very marked, most severe evidence of sign) of erythema, induration and desquamation in each of the same 4 areas. PASI score ranges from 0 (no psoriasis) to 72 (worse psoriasis). Final PASI=(sum of severity score for each area)x(% body affected score x area score).
Time Frame: Weeks 4, 8 and 12
Population: Efficacy Analysis Set (EAS) population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SRT2104 0.25 g | SRT2104 0.5 g | SRT2104 1.0 g
Number analyzed (Participants) | 7 | 9 | 12 | 11
Participants
  Week 4: 25% Improvement in PASI score from Day 1 | 2 | 1 | 3 | 7
  Week 4: 50% Improvement in PASI score from Day 1 | 0 | 0 | 1 | 0
  Week 4: 75% Improvement in PASI score from Day 1 | 0 | 0 | 0 | 0
  Week 8: 25% Improvement in PASI score from Day 1: number analyzed (Participants) | 7 | 7 | 11 | 11
  Week 8: 25% Improvement in PASI score from Day 1 | 2 | 2 | 5 | 8
  Week 8: 50% Improvement in PASI score from Day 1: number analyzed (Participants) | 7 | 7 | 11 | 11
  Week 8: 50% Improvement in PASI score from Day 1 | 1 | 2 | 4 | 4
  Week 8: 75% Improvement in PASI score from Day 1: number analyzed (Participants) | 7 | 7 | 11 | 11
  Week 8: 75% Improvement in PASI score from Day 1 | 0 | 1 | 2 | 0
  Week 12: 25% Improvement in PASI score from Day 1: number analyzed (Participants) | 7 | 6 | 9 | 11
  Week 12: 25% Improvement in PASI score from Day 1 | 2 | 2 | 6 | 8
  Week 12: 50% Improvement in PASI score from Day 1: number analyzed (Participants) | 7 | 6 | 9 | 11
  Week 12: 50% Improvement in PASI score from Day 1 | 2 | 2 | 3 | 4
  Week 12: 75% Improvement in PASI score from Day 1: number analyzed (Participants) | 7 | 6 | 9 | 11
  Week 12: 75% Improvement in PASI score from Day 1 | 1 | 2 | 2 | 1

8. Secondary Outcome: Summary of Physician's Global Assessment (PGA) Score After 4, 8 and 12 Weeks of Exposure
Description: The severity of psoriatic lesions over the whole body were assessed by the investigator using the PGA scoring system. A 0 to 6 point rating scale was used, as follows: 0 = Clear (no signs of psoriasis), 1 = Almost clear (slight elevation, scale and/or erythema), 2 = Mild (mild plaque elevation, scale and/or erythema), 3 = Mild to moderate (mild plaque elevation with moderate erythema and/or scale), 4 = Moderate (moderate plaque elevation, scale and/or erythema), 5 = Moderate to severe (marked plaque elevation, scale and/or erythema), 6 = Severe (very marked plaque elevation, scale and/or erythema). Higher scores indicated worse psoriasis. Participants in the SRT2104 0.25 g dose group inadvertently used an incorrect version of the PGA scale and thus do not have PGA data available. Participants in the SRT2104 0.25 g dose group inadvertently used an incorrect version of the PGA scale and thus do not have PGA data available.
Time Frame: Weeks 4, 8 and 12
Population: EAS Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SRT2104 0.25 g | SRT2104 0.5 g | SRT2104 1.0 g
Number analyzed (Participants) | 7 | 0 | 12 | 11
Participants
  Week 4: Very Severe: number analyzed (Participants) | 5 | 0 | 12 | 11
  Week 4: Very Severe | 1 |  | 0 | 0
  Week 4: Severe: number analyzed (Participants) | 5 | 0 | 12 | 11
  Week 4: Severe | 1 |  | 2 | 1
  Week 4: Moderate: number analyzed (Participants) | 5 | 0 | 12 | 11
  Week 4: Moderate | 2 |  | 9 | 4
  Week 4: Mild: number analyzed (Participants) | 5 | 0 | 12 | 11
  Week 4: Mild | 1 |  | 1 | 6
  Week 4: Minimal: number analyzed (Participants) | 5 | 0 | 12 | 11
  Week 4: Minimal | 0 |  | 0 | 0
  Week 4: Clear: number analyzed (Participants) | 5 | 0 | 12 | 11
  Week 4: Clear | 0 |  | 0 | 0
  Week 8: Very Severe: number analyzed (Participants) | 5 | 0 | 11 | 11
  Week 8: Very Severe | 1 |  | 0 | 0
  Week 8: Severe: number analyzed (Participants) | 5 | 0 | 11 | 11
  Week 8: Severe | 1 |  | 1 | 0
  Week 8: Moderate: number analyzed (Participants) | 5 | 0 | 11 | 11
  Week 8: Moderate | 2 |  | 6 | 3
  Week 8: Mild: number analyzed (Participants) | 5 | 0 | 11 | 11
  Week 8: Mild | 1 |  | 3 | 7
  Week 8: Minimal: number analyzed (Participants) | 5 | 0 | 11 | 11
  Week 8: Minimal | 0 |  | 1 | 1
  Week 8: Clear: number analyzed (Participants) | 5 | 0 | 11 | 11
  Week 8: Clear | 0 |  | 0 | 0
  Week 12: Very Severe: number analyzed (Participants) | 5 | 0 | 9 | 11
  Week 12: Very Severe | 1 |  | 0 | 0
  Week 12: Severe: number analyzed (Participants) | 5 | 0 | 9 | 11
  Week 12: Severe | 1 |  | 2 | 0
  Week 12: Moderate: number analyzed (Participants) | 5 | 0 | 9 | 11
  Week 12: Moderate | 2 |  | 2 | 5
  Week 12: Mild: number analyzed (Participants) | 5 | 0 | 9 | 11
  Week 12: Mild | 1 |  | 3 | 3
  Week 12: Minimal: number analyzed (Participants) | 5 | 0 | 9 | 11
  Week 12: Minimal | 0 |  | 2 | 3
  Week 12: Clear: number analyzed (Participants) | 5 | 0 | 9 | 11
  Week 12: Clear | 0 |  | 0 | 0

9. Secondary Outcome: Area Under Curve (AUC) of 12 Weeks of Dosing With 0.25 g, 0.5 g and 1.0 g SRT2104 in the Fed State in Participants
Description: A total of five blood samples (6 milliliter [mL] each) were obtained from each participant up to Week 12, for determination of SRT2104 plasma concentrations. No two samples were separated by less than an hour. One pre-dose sample was collected prior to taking study medication (30 minutes or less before dosing) at any Visit 4 (Week 4), Visit 6 (Week 8) or Visit 8 (Week 12). A single pharmacokinetic (PK) sample was collected in the time interval of 0.5 to 2 hours post-dose and also 3 to 6 hours post-dose at any Visit 4 (Week 4), Visit 6 (Week 8) or Visit 8 (Week 12). Two PK samples were collected in the time interval of 6 to 22 hours post dose at any Visit 4 (Week 4), Visit 6 (Week 8) or Visit 8 (Week 12).
Time Frame: Pre-dose (30 minutes or less before dosing: 1 sample), 0.5 to 2 hours and 3 to 6 hours post-dose (1 sample), 6 to 22 hours post-dose (2 samples) up to Week 12
Population: PK population which comprised of all participants who received at least one dose of SRT2104 for whom a PK sample was obtained and analyzed.
Measure: Mean (Standard Deviation); unit: Nanogram x hour/milliliter (ng*h/mL)
Arm/Group | SRT2104 0.25 g | SRT2104 0.5 g | SRT2104 1.0 g
Number analyzed (Participants) | 9 | 11 | 11
Nanogram x hour/milliliter (ng*h/mL) | 2148.08 (1247.182) | 4189.46 (2143.021) | 8358.45 (7466.966)

10. Secondary Outcome: Maximum Plasma Concentration (Cmax) of 12 Weeks of Dosing With 250 Milligrams (mg), 500 mg and 1000 mg SRT2104 in the Fed State in Participants
Description: A total of five blood samples (6 mL each) were obtained from each participant at any Visit 4 (Day 28 or Week 4), Visit 6 (Day 56 or Week 8) or Visit 8 (Day 84 or Week 12), for determination of SRT2104 plasma concentrations. No two samples were separated by less than an hour. One pre-dose sample was collected prior to taking study medication (30 minutes or less before dosing) at any Visit 4 (Day 28 or Week 4), Visit 6 (Day 56 or Week 8) or Visit 8 (Day 84 or Week 12). A single pharmacokinetic (PK) sample was collected in the time interval of 0.5 to 2 hours post-dose and also 3 to 6 hours post-dose at any Visit 4 (Day 28 or Week 4), Visit 6 (Day 56 or Week 8) or Visit 8 (Day 84 or Week 12). Two PK samples were collected in the time interval of 6 to 22 hours post dose at any Visit 4 (Day 28 or Week 4), Visit 6 (Day 56 or Week 8) or Visit 8 (Day 84 or Week 12).
Time Frame: One sample: Pre-dose (30 minutes or less before dosing), One sample: 0.5 to 2 hours post-dose and 3 to 6 hours post-dose and 2 samples 6 to 22 hours post dose, at any Visit 4 (Day 28 or Week 4), Visit 6 (Day 56 or Week 8) or Visit 8 (Day 84 or Week 12)
Population: PK population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SRT2104 0.25 g | SRT2104 0.5 g | SRT2104 1.0 g
Number analyzed (Participants) | 9 | 11 | 11
ng/mL | 261.64 (134.403) | 406.67 (237.787) | 1005.89 (813.346)

11. Secondary Outcome: Change From Baseline in Fibroblast Growth Factor 21 (FGF21) as an Indicator of the Pharmacodynamic Effects of SRT2104
Description: The pharmacodynamic effects of SRT2104 was measured by biomarkers of psoriatic disease activity and/or sirtuin pathway activation (hsCRP and FGF21) in blood samples. Baseline was Day 1. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values.
Time Frame: Baseline (Day 1) and Days 28, 56 and 84
Population: EAS population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picogram per milliliter
Groups:
- Placebo: Eligible participants received SRT2104 matching placebo capsules, orally, once daily after meal (at the same time every dosing day) for 84 days.
- SRT2104 0.25 g: Eligible participants received SRT2104 0.25 g capsules, orally, once daily after meal (at the same time every dosing day) for 84 days.
- SRT2104 0.5 g: Eligible participants received SRT2104 0.5 g capsules, orally, once daily after meal (at the same time every dosing day) for 84 days.
- SRT2104 1.0 g: Eligible participants received SRT2104 1.0 g capsules, orally, once daily after meal (at the same time every dosing day) for 84 days.
Arm/Group | Placebo | SRT2104 0.25 g | SRT2104 0.5 g | SRT2104 1.0 g
Number analyzed (Participants) | 7 | 9 | 12 | 11
Picogram per milliliter
  Day 28: number analyzed (Participants) | 6 | 6 | 11 | 9
  Day 28 | -61.67 (269.031) | -94.53 (154.104) | 56.93 (177.244) | 329.82 (930.329)
  Day 56: number analyzed (Participants) | 5 | 5 | 9 | 9
  Day 56 | -67.04 (276.937) | -72.72 (366.774) | 148.93 (305.634) | 268.39 (961.010)
  Day 84: number analyzed (Participants) | 5 | 4 | 9 | 9
  Day 84 | -86.12 (300.144) | -189.60 (364.475) | 58.31 (223.237) | -673.32 (1590.594)

12. Secondary Outcome: Change From Baseline in High-sensitivity C-reactive Protein (hsCRP) as an Indicator of the Pharmacodynamic Effects of SRT2104
Description: as for outcome 11
Time Frame: Baseline (Day 1) and Days 28, 56 and 84
Population: EAS population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mg per Liter
Arm/Group | Placebo | SRT2104 0.25 g | SRT2104 0.5 g | SRT2104 1.0 g
Number analyzed (Participants) | 7 | 9 | 12 | 11
mg per Liter
  Day 28: number analyzed (Participants) | 7 | 8 | 10 | 10
  Day 28 | 0.11 (2.330) | -0.14 (1.148) | 1.18 (1.954) | -0.96 (2.211)
  Day 56: number analyzed (Participants) | 7 | 6 | 7 | 10
  Day 56 | 0.59 (3.552) | -0.18 (1.897) | -1.31 (3.261) | -0.48 (2.640)
  Day 84: number analyzed (Participants) | 7 | 5 | 8 | 10
  Day 84 | 0.66 (3.895) | -0.16 (1.055) | -0.75 (3.159) | 0.27 (1.351)

ADVERSE EVENTS:
Time Frame: Up to Follow-up (Day 114)
Description: SAF Population was used.
Arm/Group | Placebo | SRT2104 0.25 g | SRT2104 0.5 g | SRT2104 1.0 g
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/9 | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/7 | 2/9 | 0/12 | 1/11
Other Adverse Events (participants affected / at risk) | 3/7 | 3/9 | 9/12 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=7) | SRT2104 0.25 g (N=9) | SRT2104 0.5 g (N=12) | SRT2104 1.0 g (N=11)
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=7) | SRT2104 0.25 g (N=9) | SRT2104 0.5 g (N=12) | SRT2104 1.0 g (N=11)
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 1
Furuncle (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Nasal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 3
Headache (Nervous system disorders) | 0 | 0 | 2 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 2
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 1
Blood potassium increased (Investigations) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Erythema annulare (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 1 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.